CLINICAL TRIAL: NCT04020367
Title: Validation of a Process for the Manufacture of Stem Cells Isolated From the Nasal Cavity for Innovative Cell Therapy of Traumatized Peripheral Nerves
Acronym: NOSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-40
Record Dates: First submitted 2019-07-11; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Septoplasty; Turbinoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with biopsy (Other)
  Interventions: Procedure: biopsy of mucosa's olfactory

INTERVENTIONS:
Procedure: biopsy of mucosa's olfactory — intervention under general or local anesthesia

SUMMARY:
Despite progress in the time taken to take charge and in the quality of the surgical technique, the repair of damaged peripheral nerves has not improved in the last twenty years. Faced with these limitations of surgical treatment, multidisciplinary teams from Marseille and Rouen have come together to propose an innovative approach to cell therapy that can limit inflammation and improve axonal growth.

Cell transplantation now appears as an alternative to treat nerve damage. Scientific advances have shown in animal models as well as in humans that mesenchymal stem cells are good cellular candidates for supporting nerve regeneration after transplantation. On the other hand, their collection requires an invasive sample most often of bone marrow. A new stem cell candidate capable of stimulating nerve regeneration has recently been identified in the olfactory mucosa located in the nasal cavity. These cells are part of the "ecto-mesenchymal" stem cell family. They have biological characteristics very similar to those of mesenchymal stem cells of the bone marrow.

They exhibit high mitogenic activity and have a high potential for differentiation towards neural lineages. Given their properties and ease of access within the nasal cavity, ecto-mesenchymal stem cells offer new perspectives for cell therapy targeting nerve damage.

In this context, nasal ecto-mesenchymal stem cells represent an interesting reconstruction alternative, particularly in the indication of peripheral nerve lesions. They are directly and easily accessible to any individual. We therefore propose in this study to validate a method of manufacturing isolated stem cells from a biopsy of a few cubic millimeters of the nasal cavity of adults, taken during a surgical procedure, with a view to proposing shortly an innovative cell therapy. From each nasal biopsy taken, the cells will be amplified in vitro under pharmaceutical grade conditions and then controlled, validated and characterized in particular for their ability to differentiate into neural cells and for their lack of genetic instability. The cells will also be cryo-preserved and then thawed under pharmaceutical grade conditions in order to validate the maintenance of their quality after cryopreservation allowing to propose a delayed implantation according to the clinical context. This study requires the taking of 25 biopsies of nasal mucosa taken from adults to document the reproducibility of the manufacturing process and possible inter-donor variations. This validation data is an essential step before considering a clinical trial of Innovative Cell Therapy Drugs.

ELIGIBILITY:
Inclusion Criteria:

* Major adults men or women
* Affiliated to a social security scheme.
* Absence of contraindication to general and / or local anesthesia
* Relevant to an operative indication of functional surgery of the nose (septoplasty and / or turbinoplasty)

Exclusion Criteria:

* Patients with proven organic pathologies of the nervous system
* Pregnant and / or lactating women
* Persons deprived of their liberty
* Major under guardianship
* persons unable to read the information document.
* Patients with chronic inflammatory and / or infectious rhinosinusitis
* Patient under antithrombotic therapy
* Patient with hypersensitivity to local amide-bound anesthetics (such as lidocaine) or to any of the components, including methyl parahydroxybenzoate contained in the vehicle.
* Patient with porphyria.
* Patient with epilepsy not controlled by treatment.
* Patient with a history of surgery on the ethmoid and / or the average turbinate bilaterally.
* Patient with a history of cervico-cephalic radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2021-02-10 (Estimated); Study Completion 2021-08-10 (Estimated)

PRIMARY OUTCOMES:
absence of caryotipic abnormalities during their amplification | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — AP-HM
Locations (1):
- Service d'Oto-Rhino-Laryngologie - Conception - AP-HM, Marseille, France